CLINICAL TRIAL: NCT05083156
Title: Cow's Milk Elimination for Treatment of Eosinophilic Esophagitis
Status: Active, not recruiting | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Joshua Wechsler, Attending Physician, Gatroenterology, Hepatology & Nutrition, Ann & Robert H Lurie Children's Hospital of Chicago
Other Study IDs: 2012-14865
Record Dates: First submitted 2021-10-06; First posted 2021-10-19 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Biospecimen Retention: Samples With DNA — 1. Intestinal Biopsies in AllProtect or RNAlater
  2. Whole Blood/Plasma/Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Milk Elimination: cohort will be observed for treatment response to elimination of cow's milk
  Interventions: Other: Diet Change

INTERVENTIONS:
Other: Diet Change — Observation Cohort will be observed for treatment response to elimination of cow's milk

SUMMARY:
The investigators seek to assess the efficacy of removing cow's milk from an EoE patient's diet. This will be determined by esophageal inflammation and clinical and histological response to the milk elimination treatment.

DETAILED DESCRIPTION:
The dietary approach is based on the hypothesis that food antigen(s) trigger eosinophilic inflammation and clinical and histological remission can be induced by identifying and excluding the causative food antigen(s). It is believed that eliminating causative food antigen(s) target the cause and thus induces long term remission.

This process is difficult as it requires multiple, invasive endoscopies and introduces the possibility of iatrogenic effects such as nutrient deficiency due to simultaneous multiple food eliminations. In addition, patient compliance may be compromised, both intentionally and unintentionally as many families report the elimination process to be both confusing and frustrating.

This prospective study eliminating only cow's milk proteins, which are a common cause of esophageal inflammation in patients with eosinophilic esophagitis, will assess the histological response in a cohort of children receiving care at Lurie Children's.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 1-18
* Patients who meet the criteria for diagnosis of EoE with ≥15 eosinophils per high power field and who had been previously treated with an adequate dose of PPI for 6-8 weeks or had a normal 24 hour ph probe study will be recruited from the patients seen by one of the physicians in the EoE clinic at Lurie Children's and other participating centers
* Patients who agree to cow's milk elimination diet as their treatment of EoE

Exclusion Criteria:

* Patients who started on oral or swallowed steroids (prior use of steroids that was discontinued more than two months prior to enrollment does not constitute an exclusion criterion)
* Patients who are unable to tolerate the cow's milk elimination diet
* Patients with concurrent eosinophilic gastroenteritis or eosinophilic colitis

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The sample size was determined based on the one-proportion non-inferiority test. The investigators recruited 54 subjects throughout the recruitment period.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Demonstrate the efficacy of the empiric single food elimination diet of eliminating cows milk | 1 year
  Participants who have eliminated cow's milk will be clinically assessed to determine if histological remission, measured by Eos/hpf, was induced under this diet for children with EOE

SECONDARY OUTCOMES:
Correlate esophageal counts with age of participant as a predictor of response | 1 year
  Participant ages will be used in statistical analysis with eosinophil counts to determine if age is a predictor of response to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Joshua B Wechsler, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H Lurie Childjren's Hospital of Chicago, Chicago, Illinois, United States